CLINICAL TRIAL: NCT00703027
Title: Diabetes Mellitus Care Decision Making Model Through Data Mining
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Principal Investigator, Ju-Ying Jiang, Attending physician, Far Eastern Memorial Hospital
Other Study IDs: 96027
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; care decision; data mining
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We tried to use data mining method to find out the new model of factors that affects the progression of diabetes mellitus.

DETAILED DESCRIPTION:
The advanced development of medical technology had led to the accumulation of a large amount of medical data. Unfortunately, these useful and meaningful clinical data were not properly managed or analyzed. Therefore, data mining technology has become an essential instrument for hospital management and medical research. Possible meaningful information can be obtained from the database through data mining. About 2,000 diabetic patients had been enrolled in Diabetes Care Program since Oct 2002 in our hospital. We intend to look for the determining factors that affect the prognosis of diabetes mellitus in our patients group.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus who had been enrolled into the Diabetes Care Program from year 2002 until 2007.

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study included 2,000 patients who visited our Division of Endocrinology and Metabolism outpatient department in this hospital with the diagnosis diabetes mellitus who had been enrolled into the Diabetes Care Program from year 2002 until 2007.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2002-10; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Ju Ying, MD, Principal Investigator — Far Eastern Memorial Hospital